CLINICAL TRIAL: NCT04365894
Title: Affective Learning in Disabled Health Training of Turkish Nursing Students: A Randomized Controlled Study
Brief Title: Affective Learning in Disabled Health Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Saglik Bilimleri University (Other)
Responsible Party: Principal Investigator, Demet İnangil, PhD, Assistant Professor, Istanbul Saglik Bilimleri University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 121234
Record Dates: First submitted 2020-04-22; First posted 2020-04-28 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Learning Disabilities
Keywords: nursing students; transformative learning; disabled
MeSH Terms: conditions — Learning Disabilities

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): The study was applied in 2nd grade nursing students' disability health course. The control group was taught with the traditional method.
- Intervention (Experimental): The intervention group with learning activities based on the transformative learning theory.
  Interventions: Other: Transformative learning theory

INTERVENTIONS:
Other: Transformative learning theory — According to the transformative learning theory, learning methods in education should include four activities as investigate, collaborative, higher-order thinking and interactive learning activities
  Arms: Intervention

SUMMARY:
This study was conducted to determine the effect of the learning method based on transformative learning theory to improve sensitivity towards the disabled on the empathic tendency, attitude and alexithymia levels of nursing students.

DETAILED DESCRIPTION:
This randomized, controlled and experimental study was conducted between October and December 2019. The sample of the study consisted of 70 2nd grade nursing students (34 people in the experimental group and 36 in the control group). The learning method based on transformative learning theory was applied to the experimental group. The data were collected using a demographic information form, the Empathic Tendency Scale, Attitudes Towards Disabled Person Scale, and Toronto Alexithymia Scale. The Mann-Whitney U Test, Wilcoxon Signed Ranks Test, Paired Sample Test, and Pearson's Chi-Squared Test were used to determine the differences between the groups.

ELIGIBILITY:
Inclusion Criteria:

* being 18 years old or above,
* to study in the second year,
* taking the theoretical course of Disabled Health

Exclusion Criteria:

* having attended any training for disabled people before
* to have any disabled person in the family members with whom they live.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
empathetic tendency | Change from baseline empathetic tendency skill at 12 weeks
  Empathetic tendency was evaluated Empathic Tendency Scale (ETS). ETS developed by Dökmen, aims to measure the potential of people to empathize in daily life. It is a five-point Likert-type scale consisting of 20 items. The responses on this scale range from "completely contradictory" to "completely eligible". While collecting points, questions 3, 6, 7, 8, 11, 12, 13, 15 are collected in reverse. The minimum score to be taken from the scale is 20, and the maximum is 100. The total scores refer to the participants' empathic tendency scores. High scores indicate high empathic tendency; low scores indicate that low empathic tendency. In the study where the scale was developed, the reliability coefficient was found to be .91.
attitude | Change from baseline attitude skill at 12 weeks
  Attitude was evaluated Attitudes Towards Disabled Person Scale (ATDPS). ATDPS was developed by Yuker and Block and adapted to Turkish by Özyürek. The aim of the scale is to measure attitudes towards people who are affected by inadequacy in general, without specifically distinguishing disability groups. This 6-point Likert-type scale consists of 20 items, which are graded as follows: "I totally agree (+3), I agree (+2), I somewhat agree (+1), I somewhat disagree (-1), I disagree (-2), I strongly disagree (-3)". Items 2, 5, 6, 11 and 12 are inverted. The sum of the points of all items is calculated, and the sign of the total score of the scale is reversed, and 60 is added to the obtained score. As a result of this calculation, the scores that can be obtained from the scale vary between 0 and 120. High scores express positive attitudes towards individuals with disabilities, and low scores mean negative attitudes.
alexithymia | Change from baseline Alexithymia skill at 12 weeks
  Alexithymia was evaluated Toronto Alexithymia Scale (TAS). This is a 20-question scale developed by Bagby et al. TAS-20 Turkish validity and reliability analyzes were performed by Gulec et al. The scale is a 5-point Likert-type measurement tool, and individuals are asked to mark the most appropriate options among "Never", "Rarely", "Sometimes", "Often" and "Always". Three sub-dimensions of the scale are difficulty identifying feelings (7 items), difficulty describing feelings (5 items) and externally oriented thinking (8 items). The reliability coefficients of the subscales are 0.82, 0.75 and 0.72, respectively. The scoring is done by summing up the points of the items. Five of these items (items 4, 5, 10, 18 and 19) are reversed. The lowest score that can be obtained from the scale is 20, and the highest score is 100. High scores indicate high alexithymia levels.

CONTACTS AND LOCATIONS:
Overall Officials: Berna Dinçer, PhD, Principal Investigator — İstanbul Medeniyet University
Locations (1):
- Saglik Bilimleri University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tsimane TA, Downing C. Transformative learning in nursing education: A concept analysis. Int J Nurs Sci. 2019 Dec 16;7(1):91-98. doi: 10.1016/j.ijnss.2019.12.006. eCollection 2020 Jan 10. PMID 32099865
- [Background] Geckil E, Kaleci E, Cingil D, Hisar F. The effect of disability empathy activity on the attitude of nursing students towards disabled people: a pilot study. Contemp Nurse. 2017 Feb;53(1):82-93. doi: 10.1080/10376178.2017.1292143. Epub 2017 Mar 2. PMID 28277092
- [Background] Seccombe JA. Attitudes towards disability in an undergraduate nursing curriculum: a literature review. Nurse Educ Today. 2007 Jul;27(5):459-65. doi: 10.1016/j.nedt.2006.08.005. Epub 2006 Oct 9. PMID 17030492